CLINICAL TRIAL: NCT04978415
Title: Comparative Study Between Peribulbar Block Technique and Sub-Tenon's Technique in Adult Patients Undergoing Redo Vitreoretinal Surgery: RCT
Brief Title: Peribulbar Block Versus Subtenon's Injection in Redo Vitreoretinal Surgery
Acronym: subtenon's
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abeer Samir Salem (Other)
Collaborators: Research Institute of Ophthalmology, Egypt (Other)
Responsible Party: Sponsor-Investigator, Abeer Samir Salem, Researcher of anesthesia, Research Institute of Ophthalmology, Egypt
Organization: Research Institute of Ophthalmology, Egypt (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: subtenon's RIO
Record Dates: First submitted 2021-07-02; First posted 2021-07-27 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- subtenon's block (Experimental): we use the subtenon cannula to inject the local anesthetic mixture
  Interventions: Procedure: peribulbar block versus subtenon's block
- peribulbar block (Experimental): we use the usual 25G sharp needle to inject the local anesthetic mixture
  Interventions: Procedure: peribulbar block versus subtenon's block

INTERVENTIONS:
Procedure: peribulbar block versus subtenon's block — Sixty patients undergoing vitreoretinal surgery were randomized to receive either peribulbar or sub-Tenon's capsule injection of 8 ml of a 20:80 mixture of 2% lidocaine and 0.75% bupivacaine with 60 IU hyalouronic acid.
  two groups 30 patient each (group p and group s) after connecting the patient to the monitor, we give him sedation 50 mg propofol, apply a nasal cannula group P: receives 2 injection peribulbar block group S: receives single injection subtenon Patients rate their pain sensation in both groups using an 11-point (0-10) numerical visual analogue scale immediately after surgery.

SUMMARY:
To compare the efficacy and efficiency of peribulbar block versus sub-Tenon's capsule injection of local anesthetic in redo vitreoretinal surgery

DETAILED DESCRIPTION:
Sixty patients undergoing vitreoretinal surgery were randomized to receive either peribulbar or sub-Tenon's capsule injection of 8 ml of a 20:80 mixture of 2% lidocaine and 0.5% bupivacaine with 60 IU hyalouronic acid.

The primary outcome measured was intraoperative eye pain, which was rated by patients in both groups using an 11-point (0-10) numerical visual analogue scale immediately after.

The surgeons indicated whether they perceived patient discomfort during 4 different stages of the operation: opening of the conjunctiva, vitrectomy (if performed), placement of scleral buckle (if performed) or using the laser probe, and closing of the conjunctiva.

The need for supplemental local anesthesia, and use of IV sedation for additional pain control intraoperatively were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80

Exclusion Criteria:

* Uncooperative patients
* Bleeding disorders
* High axial length (30mm) with previous buckle surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
intraoperative pain | during whole surgery duration (around 2 hours)
  11 point verbal rating score from 0 to 10 where 0 is no pain and 10 is intolerable pain patient will be asked immediately after surgery about pain the need for intraoperative sedation will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Samir, MD, Principal Investigator — research institute of ophthalmology
Locations (1):
- Research Institute of Ophthalmology, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided